CLINICAL TRIAL: NCT07125469
Title: Intraoperative Assessment Versus Preoperative Multidetector Computed Tomography (MDCT) for Aortic Valve Annular Sizing in Surgical Aortic Valve Replacement (SAVR)"
Brief Title: Comparing Measurements of the Aortic Valve Taken During Surgery With Those Obtained Before Surgery Using Computed Tomography Scans, in Patients Undergoing Surgical Aortic Valve Replacement
Acronym: SAVR-CT-AVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Cecilia Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SAVR-CT-AVA
Record Dates: First submitted 2025-08-05; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Valvular Heart Disease
Keywords: valve size, Surgical Aortic Valve Replacement
MeSH Terms: conditions — Heart Valve Diseases | interventions — Prostheses and Implants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with severe AS and indication to SAVR with bioprosthetic valve (Other)
  Interventions: Other: The measurements taken from the CT scan will be used to determine the appropriate size for two types of theoretical Transcatheter Aortic Valve Replacement (TAVR) prostheses

INTERVENTIONS:
Other: The measurements taken from the CT scan will be used to determine the appropriate size for two types of theoretical Transcatheter Aortic Valve Replacement (TAVR) prostheses — All patients with severe aortic stenosis (AS) who are scheduled for Surgical Aortic Valve Replacement (SAVR) with a bioprosthetic valve will undergo a pre-operative Computed Tomography (CT) scan. This CT scan will follow the pre-Transcatheter Aortic Valve Replacement (pre-TAVR) protocol and will focus only on imaging the aortic root, using a method called retrospective electrocardiogram (ECG) gating to capture detailed heart motion.
  The measurements taken from the CT scan will be used to determine the appropriate size for two types of theoretical Transcatheter Aortic Valve Replacement (TAVR) prostheses:

SUMMARY:
This study aims to understand why there may be differences between the measurements of the aortic valve taken before and during surgery. Specifically, it will compare the valve size suggested by a CT scan (Computed Tomography) with the size measured during the operation using surgical tools. This will help determine which method is more accurate for selecting the right valve size in patients undergoing SAVR (Surgical Aortic Valve Replacement ).

ELIGIBILITY:
Inclusion Criteria:

Patient age 18 years or older

All patients with isolated severe Aortic Stenosis (AS) considered eligible for Surgical Aortic Valve Replacement (SAVR) according to the current 2023 European Society of Cardiology/European Association for Cardio-Thoracic Surgery (ESC/EACTS) guidelines for management of Valvular Heart Disease (reference 8) will be enrolled.

Patient is willing to comply with study procedures and is available to return to the center for follow-up visits.

Informed consent documentation signed and dated confirming that the patient has been adequately informed of all aspects related to his/her participation in the clinical study and is willing to participate.

Exclusion Criteria:

Bicuspid aortic valve anatomy Moderate to severe aortic valve regurgitation Multivalvular disease Redo Surgical Aortic Valve Replacement Ascending aorta aneurysm Aortic root enlargement Chronic Kidney Disease with estimated Glomerular Filtration Rate less than 30 milliliters per minute Body Mass Index greater than 30 kilograms per square meter Inadequate Multidetector Computed Tomography images

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Aortic Valve Annular sizing in Surgical Aortic Valve Replacement | pre-operative
  All patients with severe aortic stenosis (narrowing of the aortic valve) scheduled for Surgical Aortic Valve Replacement (SAVR), which is open-heart surgery to replace the valve with a bioprosthetic (tissue) valve, will have a pre-operative Computed Tomography (CT) scan. This CT scan follows the pre-Transcatheter Aortic Valve Replacement (pre-TAVR) protocol and focuses on the aortic root (the base of the aorta). It uses retrospective electrocardiogram (ECG) gating, a technique that times image capture with the heartbeat to get clear pictures of the heart.

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Castriota, Principal Investigator — Maria Cecilia Hospital
Locations (1):
- Maria Cecilia Hospital, Cotignola, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared. However, de-identified data may be made available to qualified researchers upon reasonable request to the study center and the Principal Investigator. All data will be processed in compliance with the General Data Protection Regulation (GDPR - EU Regulation 2016/679), ensuring the confidentiality, integrity, and protection of participants' personal information.